CLINICAL TRIAL: NCT04398407
Title: Testing the Effectiveness of Mainstream Management Tools to Increase Organizational Commitment and Job Satisfaction and Decrease Turnover Among Peer Providers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5348E
Record Dates: First submitted 2020-05-14; First posted 2020-05-21 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Mental Health; Work Related Stress
Keywords: peer support specialists; coaching
MeSH Terms: conditions — Psychological Well-Being; Occupational Stress

STUDY DESIGN:
Intervention Model Description: This study in a randomized control trial, with an enhanced control condition. Prior to the randomized trial, the investigators will conduct a small pilot study. Findings from the pilot study will inform revisions of the intervention prior to the randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching and Achievement of Peer Providers (CAPP) (Experimental): CAPP will consist of 16 individualized, one-on-one sessions using Zoom or other videoconferencing software and occurring over a 4-month period. Coaching meetings will take approximately one hour per week. The coach will tailor and individualize the modules and time spent on modules to meet the goals of each peer provider.
  Modules:
  Module 1: Establishing and solidifying the working alliance, understanding the work setting and role Module 2: Understand Generic drivers of burnout and role stress Module 3: Discuss specific sources of role stressors and burnout Module 4: Set SMART Goals Module 5: Overcome challenges for workplace success Module 6: Develop Skills for Workplace Success Module 7: Managing co-worker and supervisory relations in the workplace Module 8: Wrap-up sessions
  During the first stage of research, the CAPP intervention will be further developed and refined, prior to the Randomized clinical trial.
  Interventions: Behavioral: Coaching and Advancement for Peer Providers (CAPP)
- Enhanced control (Active Comparator): The "enhanced" control condition will include 1 generic informational session conducted by a CAPP coach.During that session, the coach will introduce the key concepts under study and provide information about the drivers of burnout and role stress. The CAPP coach will discuss the need to set goals to overcome these challenges and will provide one article via email describing burnout and role stressors that is suitable for a lay person.
  Interventions: Behavioral: Coaching and Advancement for Peer Providers (CAPP)

INTERVENTIONS:
Behavioral: Coaching and Advancement for Peer Providers (CAPP) — The CAPP intervention will combine executive coaching approaches and techniques with the specific needs and environmental demands of individuals working as PSS. A person who has been a PSS and trainer of PSS nationally has developed the CAPP intervention using the expertise of Center staff, the Harvard Institute of Coaching (IOC) and our Peer Advisory Group. Individuals randomized to the experimental condition will receive 16 individual coaching sessions tailored to the specific job stressors they are experiencing. CAPP is designed to address the following issues: role confusion, lack of clarity about job tasks, conflict with other providers, burnout, lack of organizational commitment and job satisfaction.

SUMMARY:
The role of peer support specialists (PSS) has burgeoned in the mental health field. Peer support specialists are individuals with a psychiatric condition who are in recovery and who are employed to provide various kinds of tangible and other supports to individuals with psychiatric conditions, generally in public mental health programs. Partially because of the newness of this role, PSS experience confusion about their role and tasks as well as conflict with other mental health providers who are uncertain about how to utilize PSS effectively in services.

This project was designed to bring a coaching service to PSS to assist them to address challenges in their job. The investigators will conduct a randomized control trial to evaluate a novel coaching, Coaching and Advancement for Peer Providers (CAPP). Our hypotheses are that individuals participating in the CAPP intervention will experience a reduction in burnout, role confusion, and intention to leave their job or the field. Participants in CAPP will also experience an increase in job satisfaction, role clarity and organizational commitment.

DETAILED DESCRIPTION:
The role of peer support specialists (PSS) has burgeoned in the mental health field. Peer support specialists are individuals with a psychiatric condition who are in recovery and who are employed to provide various kinds of tangible and other supports to individuals with psychiatric conditions, generally in public mental health programs. Partially because of the newness of this role, PSS experience confusion about their role and tasks as well as conflict with other mental health providers who are uncertain about how to utilize PSS effectively in services.

This project was designed to bring a coaching service to PSS to assist them to address challenges in their job. There are three phases of this study:

1. The investigators will test components of the intervention with volunteers who are peer specialists. The investigators will collect no data from these individuals and will use the information gathered to refine the intervention.
2. Next, the investigators will recruit and randomly assign 140 PSS to participate in this newly developed coaching intervention (Coaching and Advancement for Peer Providers, or CAPP) and to assess their level of role confusion, overload, burnout, and intention to leave their job or their profession.
3. Finally, the investigators will conduct a qualitative study of experimental study participants to learn about the experience of CAPP.

Individuals will be randomly assigned to receive CAPP or an informational control group. A total of 16 CAPP sessions will be conducted with coaches that the investigators train and supervise. This will be a telehealth intervention and study. That is, all consenting and coaching sessions will be conducted using platforms such as Zoom (HIPAA compliant version) and assessments will be collected using online platforms (REDCap). Individuals will be assessed at baseline, 4, 6, and 9 months after baseline. The investigators will record selected coaching sessions to insure that the intervention is being delivered with fidelity. Our hypotheses are that individuals participating in the CAPP intervention will experience a reduction in burnout, role confusion, and intention to leave their job or the field. Participants in CAPP will also experience an increase in job satisfaction, role clarity and organizational commitment.

ELIGIBILITY:
Inclusion Criteria:

Peer support specialists/providers who are:

1. are currently employed a minimum of 10 hours per week as an employee in a mental health setting;
2. are providing services to individuals with psychiatric disabilities (this will exclude individuals in volunteer positions);
3. have been employed as a peer provider for a minimum of 6 months;
4. are employed in a mental health program;
5. express types of concerns about their work, such as distress or lack of clarity about their job, role stressors and/or burnout, that suggest they could benefit from the intervention;
6. express a willingness to engage in the CAPP Coaching intervention;
7. have the ability to conduct CAPP sessions and assessments in English.

Exclusion Criteria:

1. unable or unwilling to provide full and knowing consent for the research study;
2. unwilling to participate in the data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Effort-Reward Imbalance Scale-assessing change | Baseline, immediately after the intervention, 6 months followup, 9 months followup
  Examines role over load and related concepts, including role ambiguity, role conflict, and role overload. Range: 16-64, higher values indicate higher imbalance.
Utrecht Work Engagement Scale-Short Form-assessing change | Baseline, immediately after the intervention, 6 months followup, 9 months followup
  Measures engagement in one's work. The scale measures vigor, dedication and absorption at work. Items include "I am proud of the work I do" and "I am immersed in my work". Respondents answer on a 7-point scale ranging from Never to Always.
Quality of Work Life (QWL)-assessing change | Baseline, immediately after the intervention, 6 months followup, 9 months followup
  Select items from the QWL. The QWL captures many aspects of work life; including various aspects of Work Climate, such as: Safety, Discrimination, Harassment, Respect, Trust, and Management Relationship. Example items include: "My supervisor is concerned with the welfare of those under him or her," "The people I work with take a personal interest in me." Items are rated on a 4-point Likert scale from "Not at all true" to "Very True." National Opinion Research Center reports excellent psychometric properties of the scale. This scale will be primarily used to examine organizational/work climate.
Job satisfaction-assessing change | Baseline, immediately after the intervention, 6 months followup, 9 months followup
  Job Satisfaction will be assessed using the items validated by Lee and his colleagues (Lee, et al., 2018). This measure is designed to assess global job satisfaction and appraisal of one's job responsibilities. Sample items include: "Generally speaking, I am very satisfied with this job" and "I am generally satisfied with the kind of work I do in this job." To assess global job satisfaction, one item from the Michigan Organizational Assessment Questionnaire (MOAQ) ("All in all I am satisfied with my current job") will also be administered.
Turnover intention-assessing change | Baseline, immediately after the intervention, 6 months followup, 9 months followup
  Three items from the Intention-to-Leave scale (XXX & Levin, 2006) e.g., "In the next few months I intend to leave this organization" will be used to capture turnover intention. Items are rated on a 7-point, Likert-type scale ranging from "Strongly Disagree" (1) to "Strongly Agree" (7).
  In addition, the investigators will also examine actual job turnover at all assessment time periods.
Goal Attainment Scaling-assessing change | Baseline, immediately after the intervention, 6 months followup, 9 months followup
  Goal Attainment Scale provides a structured approach to determining goal achievement regardless of the type or uniqueness of goal. As part of the intervention, individuals will be asked to set two work related goals (from a preestablished list of goals) that addresses their source of distress. At followup, participants will be asked to assess their progress using the Goal Attainment Scale (-2: much lower than expected; 0: expected goal achievement; +2: much higher than expected).
Maslach Burnout Inventory-Human Services Survey-assessing change | Baseline, immediately after the intervention, 6 months followup, 9 months followup
  This scale assesses multiple facets of burnout: emotional exhaustion, depersonalization, and sense of personal accomplishment. Items are rated based on frequency of their occurrence from "Never" to "Every Day" and include: "I feel emotionally drained from my work," "I have accomplished many worthwhile things in this job," "I don't really care what happens to some recipients." Scores range from 0-132, with high scores indicating higher burnout.
Three Component Organizational Commitment Scale-assessing change | Baseline, immediately after the intervention, 6 months followup, 9 months followup
  The three component organization commitment scale evaluates affective, continuance, and normative commitment to an organization. Affective components assess the desire of an employee to remain with an organization ("I would be very happy to spend the rest of my career with this organization") while continuance commitment assesses the person's need to remain with the organization ("It would be very hard for me to leave my organization right now, even if I wanted to"). Finally, normative commitment assesses the person feeling that they should remain with the organization ("I think that people these days move from company to company too often"). Items are measured on a 7-point scale from Strongly Disagree to Strongly Agree.

OTHER OUTCOMES:
Working alliance inventory | Immediately after the intervention for experimental condition only
  12-item instrument that provides information about the extent to which a provider and recipient, a) share mutual goals (e.g., "__[coach name]__ and I are working towards mutually agreed upon goals"), b) agree on tasks needed to accomplish those goals (e.g., "We have established a good understanding of the kind of changes that would be good for me"), and c) have developed a bond (e.g., "I feel that __[coach name]__ appreciates me") using a 7-point scale ranging from Always to Never.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided